CLINICAL TRIAL: NCT02060838
Title: The Impact of Storage Techniques on Platelets Number and Function After Acute Normovolemic Hemodilution (ANH)
Status: Completed | Type: Observational
Sponsor: Aymen N Naguib (Other)
Responsible Party: Sponsor-Investigator, Aymen N Naguib, Director of Pediatric Cardiothoracic Anesthesia, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00762
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2016-10

CONDITIONS: Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute normovolemic hemodilution (ANH): Patients undergoing acute normovolemic hemodilution (ANH) as part of their cardiac surgery.
  Interventions: Procedure: Acute normovolemic hemodilution (ANH)

INTERVENTIONS:
Procedure: Acute normovolemic hemodilution (ANH) — Blood is drawn from our patients pre-bypass after obtaining the arterial line and administered back to the patient after separation from cardiopulmonary bypass (CPB) and reversal of heparin with protamine.

SUMMARY:
Acute normovolemic hemodilution (ANH) is part of our current protocol to decrease post-operative bleeding and homologous blood transfusions post cardiopulmonary bypass. Blood is drawn from our patients pre-bypass after obtaining the arterial line and administered back to the patient after separation from cardiopulmonary bypass (CPB) and reversal of heparin with protamine. In our practice we noticed some variability in the impact of ANH on postoperative bleeding; with some patients appearing to show more hemostasis after separation from CPB than others. This is a prospective study to find out if there is an optimal time period that guarantees the largest amount of functioning platelets and what is the best practice for drawing and storing of ANH to guarantee the largest amount of functioning platelets.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing cardiac surgery on CPB and are determined to be suitable for ANH by the cardiac team during the huddle process per our standard protocol.

Exclusion Criteria:

* Patients who are undergoing cardiac surgery on CPB who are determined not to be suitable candidates for ANH by the cardiac team during the huddle process per our standard protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing open-heart surgery who will be having acute normovolemic hemodilution (ANH) as part of their surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Result] Sebastian R, Ratliff T, Winch PD, Tumin D, Gomez D, Tobias J, Galantowicz M, Naguib AN. Revisiting acute normovolemic hemodilution and blood transfusion during pediatric cardiac surgery: a prospective observational study. Paediatr Anaesth. 2017 Jan;27(1):85-90. doi: 10.1111/pan.13014. Epub 2016 Oct 13. PMID 27734554

RESULTS

PARTICIPANT FLOW:
Groups:
- ANH Collected & Stored in a Bag; ANH Collected & Stored in a Syringe: Patients undergoing acute normovolemic hemodilution (ANH) as part of their cardiac surgery.
  Acute normovolemic hemodilution (ANH): Blood is drawn from our patients pre-bypass after obtaining the arterial line and administered back to the patient after separation from cardiopulmonary bypass (CPB) and reversal of heparin with protamine.
Period: Overall Study
Arm/Group | ANH Collected & Stored in a Bag | ANH Collected & Stored in a Syringe
Started | 28 | 22
Completed | 28 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ANH Blood Collected in a Bag: Patients undergoing acute normovolemic hemodilution (ANH) as part of their cardiac surgery.
  Acute normovolemic hemodilution (ANH): Blood is drawn from our patients pre-bypass after obtaining the arterial line, stored in an IV infusion bag, and administered back to the patient after separation from cardiopulmonary bypass (CPB) and reversal of heparin with protamine.
- ANH Blood Collected in a Syringe: Patients undergoing acute normovolemic hemodilution (ANH) as part of their cardiac surgery.
  Acute normovolemic hemodilution (ANH): Blood is drawn from our patients pre-bypass after obtaining the arterial line, stored in a syringe, and administered back to the patient after separation from cardiopulmonary bypass (CPB) and reversal of heparin with protamine.
- Total: Total of all reporting groups
Arm/Group | ANH Blood Collected in a Bag | ANH Blood Collected in a Syringe | Total
Number analyzed (Participants) | 28 | 22 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 22 | 41
  Between 18 and 65 years | 9 | 0 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14.6 [11.0 to 20.8] | 3.0 [1.0 to 5.7] | 8.3 [3.1 to 15.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 20 | 13 | 33

OUTCOME MEASURES:

1. Primary Outcome: Time to Platelet Aggregation as Measured Using Collagen-epinephrine (EPI)
Description: The membrane of the cartridges are coated with collagen and epinephrine (EPI) inducing a platelet plug to form which closes the aperture.
Time Frame: Just prior to re-transfusion, assessed up to 5 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | ANH Blood Collected in a Bag | ANH Blood Collected in a Syringe
Number analyzed (Participants) | 28 | 22
seconds | 260 [234 to 282] | 261 [233 to 283]

2. Primary Outcome: Time to Platelet Aggregation as Measured Using Collagen-Adenosine (ADP)
Description: The membrane of the cartridges are coated with collagen and adenosine diphosphate (ADP) inducing a platelet plug to form which closes the aperture.
Time Frame: Just prior to re-transfusion, assessed up to 5 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | ANH Blood Collected in a Bag | ANH Blood Collected in a Syringe
Number analyzed (Participants) | 28 | 22
seconds | 251 [221 to 267] | 245 [225 to 295]

ADVERSE EVENTS:
Groups:
- ANH Blood Collected & Stored in a Bag: Patients undergoing acute normovolemic hemodilution (ANH) as part of their cardiac surgery.
  Acute normovolemic hemodilution (ANH): Blood is drawn from our patients pre-bypass after obtaining the arterial line, stored in an IV infusion bag, and administered back to the patient after separation from cardiopulmonary bypass (CPB) and reversal of heparin with protamine.
- ANH Blood Collected & Stored in a Syringe: Patients undergoing acute normovolemic hemodilution (ANH) as part of their cardiac surgery.
  Acute normovolemic hemodilution (ANH): Blood is drawn from our patients pre-bypass after obtaining the arterial line, stored in a syringe, and administered back to the patient after separation from cardiopulmonary bypass (CPB) and reversal of heparin with protamine.
Arm/Group | ANH Blood Collected & Stored in a Bag | ANH Blood Collected & Stored in a Syringe
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/22
Other Adverse Events (participants affected / at risk) | 0/28 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes